CLINICAL TRIAL: NCT03036046
Title: An Open Label Phase IIa Clinical Study to Evaluate the Safety and Pharmacokinetics of Oral F901318 (Combined With Fluconazole and Posaconazole) in AML
Brief Title: Safety and Pharmacokinetics of Oral F901318 (Fluconazole and Posaconazole) IN Aml Leukaemia
Acronym: SAFEGUARDFP
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study no longer required
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: The Clinical Trials Centre Cologne (Other); Klinik für Hämatologie, Aachen (Unknown); Medizinische Klinik Würzburg (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F901318C21
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — olorofim; Fluconazole; posaconazole

STUDY DESIGN:
Intervention Model Description: Patients in group low dose fluconazole will be enrolled ahead of group high dose fluconazole. Group posaconazole will be enrolled in parallel according to prevaling practice in the institutions involved in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- F901318 with fluconazole low dose (Experimental): safety assessment
  Interventions: Drug: F901318 with fluconazole low dose
- F901318 with fluconazole high dose (Experimental): safety assessment
  Interventions: Drug: F901318 with fluconazole high dose
- F901318 with posaconazole (Experimental): safety assessment
  Interventions: Drug: F901318 with posaconazole

INTERVENTIONS:
Drug: F901318 with fluconazole low dose — adverse events
  Arms: F901318 with fluconazole low dose
Drug: F901318 with fluconazole high dose — adverse events
  Arms: F901318 with fluconazole high dose
Drug: F901318 with posaconazole — adverse events
  Arms: F901318 with posaconazole

SUMMARY:
Non-randomized, multi-centre, open label, uncontrolled, multiple dose, phase IIa study.

A total of 18 patients diagnosed with acute myeloid leukaemia (AML) scheduled for chemotherapy and expected to be neutropenic (<500 Absolute neutrophil count (ANC)/µl) for >10 days will be treated. F901318 will be given in conjunction with fluconazole or posaconzaole in order to assess safe treatment regimens for both combinations.

DETAILED DESCRIPTION:
'F901318 has potent in vitro efficacy against Aspergillus spp. including azole-resistant strains and consistent efficacy in in vivo mouse models of infection. F901318 is active by both oral and intravenous routes of administration in preclinical efficacy studies.

Non-clinical studies and phase I clinical trials show that F901318 has a good overall safety profile and limited potential for drug-drug interactions. F901318 exhibits a highly promising profile which can potentially address the critical treatment requirements for invasive Aspergillus infections in a changing clinical environment in which new classes of antifungals are needed.

This phase IIa study aims to confirm PK and safety information of F901318 from phase I and bridge them to a neutropenic AML patient population, which represents the main population for future efficacy trials. Coadministration of fluconazole or posaconazole will allow recognizing potential factors of suboptimal F901318 exposure without the risk of fatal disseminating infection.'

ELIGIBILITY:
Inclusion Criteria:

* Participating patients need to fulfil all of the following criteria:

  1. Patients diagnosed with AML and entering treatment of chemotherapy.
  2. Patients are expected to be neutropenic (ANC <500/µl) for >10 days.
  3. Provision of written informed consent prior to any study specific procedures.
  4. Ability and willingness to comply with the protocol.
  5. Patients aged over 18 years.
  6. Patients with body weight ≥60 kg
  7. Group F only: patient receives according to local clinical standard either

     * no fungal prophylaxis or
     * only topical fungal prophylaxis (e.g. Ampho moronal®) or
     * fluconazole as routine fungal prophylaxis
  8. Group P only: patient receives posaconazole as fungal prophylaxis according to local clinical standard

Exclusion Criteria:

* Any of the following will exclude a patient from the study:

  1. Documented lung infiltrate at screening.
  2. Evidence for active fungal infection, such as documented serum GMI ≥0.5 at screening (within 5 days before study start)
  3. Current IFD or prior history of IFD or patients who received systemic antifungal therapy for proven or probable IFD in the last 12 months.
  4. Patients who received any systemic antifungal therapy for more than 72 hours immediately prior to first administration of study medication. Echinocandins, posaconazole (group P, see also inclusion criterion 8), and topical polyenes or nystatin are acceptable.
  5. Concomitant exposure to phenobarbital and long acting barbiturates, triazolam, carbamazepine, phenytoin, pimozide, cisaprid, efavirenz, ritonavir, rifabutin, rifampicin, ergot alkaloids (ergotamine, dihydroergotamin), ibrutinib, idelalisib, vinca alkaloids, digoxin, dofetilide, quinidine, St. John´s wort, everolimus, sirolimus, astemizole, terfenadine, methadone, alfentanil, fentanyl and other structurally related opiates, warfarin (see also section 8.8 for details).
  6. Documented prolongation of the QTc interval (>450 ms).
  7. Concomitant medication that prolongs QT interval (except for cytostatic drugs used during chemotherapy, such as mitoxantrone).
  8. Any other concomitant medical condition that, in the opinion of the investigator, may be an unacceptable additional risk to the patient should he/she participate in the study.
  9. History of convulsion.
  10. Female patients only: Positive result of pregnancy test or breastfeeding.
  11. Female patients of childbearing potential who do not practice sexual abstinence as their common way of life and confirm to stay sexually abstinent also during their participation in the study or who do not use or do not agree to use appropriate contraceptive methods (prior to and during the study, including 14 days after the last dose of study therapy) as defined in ICH guideline M3(R2) on non-clinical safety studies for the conduct of human clinical trials and marketing authorisation for pharmaceuticals (EMA/CPMP/ICH/286/1995). Hormonal contraception alone is not considered appropriate. See section 9.3.2 for additional information.
  12. Known hypersensitivity to any component of the study medication.
  13. A history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalaemia, cardiomyopathy, sinus bradycardia, symptomatic arrhythmias, family history of long QT Syndrome).
  14. Patient has had acute hepatitis in the prior 6 months, chronic hepatitis, cirrhosis (any Child-Pugh class), acute hepatic failure, or acute decompensation of chronic hepatic failure
  15. Presence of hepatic disease as indicated by aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 × upper limit of normal (ULN) at Screening. Patients with AST and/or ALT >3 × ULN and <5 × ULN are eligible if these elevations are acute, not accompanied by a total bilirubin ≥2xULN and documented by the investigator as being directly related to an infectious process being treated. During the clinical study, the investigator is responsible for, without delay, determining whether the patient meets potential Hy's law criteria (according to FDA [16]).
  16. Patient has a total bilirubin >3 × ULN, unless isolated hyperbilirubinemia is directly related to an acute infection or due to known Gilbert's disease.
  17. Calculated creatinine clearance (CrCl) <50 mL/minute.
  18. Medical history of oliguria (<20 mL/h) unresponsive to fluid challenge.
  19. Suspected other or additional cause for neutropenia or immunosuppression (other than AML or myelodysplastic syndrome).
  20. Any other medical condition, which may affect the clinical evaluability of the patient.
  21. Patients previously enrolled in this study.
  22. Patient has participated or intends to participate in any other clinical study that involves the administration of an investigational medication at the time of presentation, during the course of the study, or during the 30 days prior to study start. New combinations of labelled substances for chemotherapy are allowed.
  23. Chronic external ocular disease
  24. Contact lens use intended during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | 63 days
  Adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (Area under concentration/time curve) | 14 days
  Area under concentration/time curve

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A Cornely, MD, Principal Investigator — University Hospital Cologne

IPD SHARING:
Plan to Share IPD: No